CLINICAL TRIAL: NCT03711825
Title: An Open Label Study to Evaluate the Safety and Gastric-Retentive Properties of Modified Release Capsules Containing Memantine Hydrochloride in Healthy Adults
Brief Title: Study to Evaluate Safety/Duration in Stomach of Extended Release Capsules Containing Memantine Hydrochloride in Healthy Adults
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Lyndra Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LYN-057-C-002; ACTRN12618001426279 (Registry Identifier: ANZCTR); CM8718 (Other: CMAX)
Record Dates: First submitted 2018-10-14; First posted 2018-10-19 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Alzheimer Disease; Gastric Retention; Healthy
MeSH Terms: conditions — Alzheimer Disease | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sentinel/Main (Experimental): Sentinel dosing of two subjects in clinic of LYN-057 (50 mg), followed by Main, i.e. remaining 6 subjects, for total of 8 subjects doses; followed by imaging assessment (MRI/abdominal U/S)
  Interventions: Drug: LYN-057; Procedure: Imaging Assessment (MRI); Procedure: Imaging Assessment (U/S)

INTERVENTIONS:
Drug: LYN-057 — Administration of single dose of LYN-057 presented as extended release capsule containing 50 mg of memantine hydrochloride (HCl)
  Other Names: LYN-057 (50 mg)
Procedure: Imaging Assessment (MRI) — Imaging assessments [MRI] will be performed on specified days according to protocol
  Other Names: MRI
Procedure: Imaging Assessment (U/S) — Imaging assessments (abdominal U/S) will be performed on specified days according to protocol
  Other Names: Abdominal Ultrasound

SUMMARY:
To assess how long memantine hydrochloride (HCl) (50 mg) extended release capsules stay in the stomach as determined by imaging assessment (MRI or abdominal ultrasound).

To evaluate the safety of a memantine HCl extended release capsule formulation

DETAILED DESCRIPTION:
This is a single centre, open label, single dose study in healthy adult subjects.

Eligible individuals will be admitted to an inpatient unit in two or more cohorts. Enough eligible individuals will be admitted allowing for the enrollment of the Sentinel (n= 2) and Main Group (total of n=8 in Main), and an optional Supplemental Group (n= 6), if required.

All enrolled subjects will be dosed with a single administration of an extended release capsule containing memantine hydrochloride (LYN-057), 50 mg. Dosing will be conducted in an inpatient clinical unit, with access to an acute care facility. Subjects will remain in the inpatient unit for 7 days after dosing. During this time, subjects will undergo intermittent imaging assessments for gastric retention [magnetic resonance imaging (MRI) and abdominal ultrasound (U/S)], safety assessments, blood sampling for evaluation of memantine pharmacokinetics (PK), and faecal collections for assessments of formulation components and bowel movement characteristics.

Subjects will return to the clinic for PK sampling and safety assessments on Days 10, 15, 22 and Day 29 (End of Study Visit). In addition, some subjects may continue to perform faecal collection and/or may undergo imaging assessments on Day 10 based on clinical criteria. On Day 29 (End of Study Visit), subjects will undergo final safety and PK assessments and will be discharged from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects
2. Body mass index of 18.0 to 30.0 kg/meters-squared
3. Suitable scores for two swallowing questionnaires
4. Demonstrate normal swallowing and gastrointestinal passage for capsule, as assessed while undergoing imaging studies
5. Must provide written informed consent

Exclusion Criteria:

1. Participants who have previously been enrolled in this study
2. History of any drug or alcohol abuse in the past 2 years
3. Current smokers and those who have smoked within the past 12 months
4. Individuals with clinically significant medical history relating to the gastrointestinal tract and potential complications, thereof
5. Individuals with a positive test for HIV, hepatitis B or hepatitis C
6. Individuals who are contraindicated based on memantine HCl
7. Serious adverse reaction or serious hypersensitivity to components of the study formulation or patency capsule
8. Individuals who have received any experimental agent within 30 days (or 5 half-lives), whichever is longer, prior to the date of dosing
9. Individuals with contraindication to MRI imaging
10. Individuals with functional constipation, irritable bowel, or functional diarrhea, as evaluated by standardized questionnaire
11. Individuals with contraindications to elective X-ray based on known or expected radiation exposure

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-11-13 (Actual)

PRIMARY OUTCOMES:
Gastric retention by imaging assessment by MRI | Up to 9 days post-dosing
  Visualization of formulation/formulation components in stomach by MRI
Gastric retention by imaging assessment by abdominal U/S | Up to 9 days post-dosing
  Visualization of formulation/formulation components in stomach by abdominal U/S
Safety and tolerability of a single dose of LYN-057 extended release capsule | Through study completion, up to 3 months
  Safety collected from a combination of the following: Adverse Event (AE) reporting and examinations specified per protocol

SECONDARY OUTCOMES:
Memantine HCl pharmacokinetics - Maximum Plasma Concentration (Cmax) | Pre-dose, on day of dosing at 2, 4, 6, 8 and 12 hours post-dosing, thereafter daily during inpatient stay through Day 8. After Day 8, PK sampling on Day 10, 15, 22 and 29.
  Memantine HCl pharmacokinetics - Cmax by validated assay
Memantine HCl pharmacokinetics - Time after administration of maximum plasma concentration (Tmax) | Pre-dose, on day of dosing at 2, 4, 6, 8 and 12 hours post-dosing, thereafter daily during inpatient stay through Day 8. After Day 8, PK sampling on Day 10, 15, 22 and 29.
  Memantine HCl pharmacokinetics - Tmax by validated assay
Memantine HCl pharmacokinetics - Area Under the Curve (AUC) | Pre-dose, on day of dosing at 2, 4, 6, 8 and 12 hours post-dosing, thereafter daily during inpatient stay through Day 8. After Day 8, PK sampling on Day 10, 15, 22 and 29.
  Memantine HCl pharmacokinetics - AUC by validated assay
Physical features of recovered formulation components | Through study completion, up to 29 days
  Recording of the descriptive physical features, e.g. number of polymeric arms (if separate) or attached to the core, of formulation components recovered from collected fecal specimens

CONTACTS AND LOCATIONS:
Overall Officials: Sepehr Shakib, MD, Principal Investigator — CMAX
Locations (1):
- CMAX, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No